CLINICAL TRIAL: NCT03706950
Title: Multicentre, Open-label, Post-approval Observational Study of Elpida® Used in the First Line Therapy for HIV-1 Infected Patients With the Background of Standard Baseline ART (NNRTI + 2 NRTIs)
Brief Title: Post-approval Observational Study of Elpida® in the First Line Therapy for HIV-1 Infected Patients With Background Standard ART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Other Study IDs: HIV-VM1500-06
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: HIV-1-infection
Keywords: HIV-1
MeSH Terms: interventions — elsulfavirine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elpida® + 2 NRTIs: Elpida® 20mg qd in the first line of therapy for HIV-1 infected patients with a background standard ART.
  Interventions: Drug: Elpida® + 2 NRTIs

INTERVENTIONS:
Drug: Elpida® + 2 NRTIs — Elpida® 20mg qd orally + 2 NRTIs standard prescribed ART therapy

SUMMARY:
This post-registration observational study is designed to monitor the safety parameters and efficacy of Elpida® in actual practice in the first-line treatment of HIV-1 infected patients on the background of the standard baseline ART.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, post-registration observational non-interventional study of the use of Elpida® in the first line of therapy for HIV-1 infected patients against a background of standard baseline ART (NNRTIs + 2 NRTIs). The study is scheduled to be conducted approximately in 20 centers for the prevention and control of AIDS in Russia.

In total, 2000 HIV-1-infected patients who are prescribed therapy with Elpida® (20 mg capsules) against the background of standard baseline ART are planned to be included in the study.

The observational study will collect data from patients who signed informed consent and meet all inclusion/non-inclusion criteria from the time that precedes the therapy by Elpida® up to 96 weeks of treatment or until early elimination. The data will be obtained through routine visits and procedures, including demographics and history, height, body weight, body mass index (BMI), laboratory data (viral load of HIV-1, CD4+-T-lymphocytes, resistance mutations in HIV-1, screening for hepatitis B and C, syphilis, general and biochemical blood analysis, general urine analysis) and instrumental examinations (electrocardiography (ECG), chest X-ray/fluorography). Throughout the study, patients will keep observation diaries for recording AEs and concomitant therapy. Data on the intake of ART drugs and AE related to their use will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. A signed patient information sheet and a form of informed consent to participate in the study.
2. Men and women aged 18 and over.
3. Document supported HIV-1 infection.
4. Patients whom during the previous 24 weeks first line ART was prescried comprising the drug Elpida®, including patients who are ART-naive or were transferred to Elpida® from other first line ART regimens due to intolerance (transfer from other NNRTIs - within the class; transfer from protease inhibitors, including boosted ones, due to lipid metabolism disorders or other adverse reactions (AR) if the virological effectiveness of the previous ART regimen - was effective - reaching undetectable levels of viral load).

Exclusion Criteria:

1. Current participation in the clinical trial.
2. Significant alcohol and/(or) drug dependence, which, according to the researcher, can prevent collection of data.
3. Increase of AST/ALT levels by more than 2.5 times higher than the upper limit of the reference range at Week 0 visit.
4. Replication stage of chronic hepatitis C (presence of HCV RNA), requiring therapy.
5. Use of Elpida® in violation of indications officially approved by the Ministry of Health of the Russian Federation on the package leaflet.
6. Significant secondary diseases requiring treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In total, 2000 HIV-1-infected patients who are prescribed therapy with Elpida® (20 mg capsules) against the background of standard baseline ART are planned to be included in the observational study. The study will enroll patients who are ART-naive or are transferred to Elpida® from other first-line ART regimens because of intolerance.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs | 96 weeks
  Incidence of adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Viral load | 96 weeks
  Dynamics of viral load (HIV RNA) in blood plasma
Proportion of patients with undetectable viral load on visits, starting from Week 24 | 24 weeks
  Proportion of patients with undetectable viral load (HIV-1 RNA level in blood plasma < 50 copies / ml or, at least 400 copies / ml depending on assessment method sensitivity in the clinical site) on visits, starting from Week 24
The frequency of virological failures | 96 weks
  The frequency of virological failures, including incomplete suppression or the resumption of viral load
Absolute CD8+ lymphocytes count | 96 weeks
  Change in the absolute CD8+ lymphocytes count
The percent of patients who developed HIV-1 resistance to Elpida® | 96 weeks
  The proportion of patients who develop study therapy-resistant HIV-1. An assessment of the development of HIV-1 resistance to antiretroviral drugs should be carried out if treatment failure is registered. Treatment failure is determined after at least 24 weeks of therapy, if in two consecutive measurements with an interval of 12 weeks the viral load exceeds 1000 copies / ml providing patient complience with ART recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Elena Yakubova, PhD, Study Director — Viriom
Locations (11):
- Russia (11):
  - Regional AIDS Prevention and Control Center, Astrakhan
  - Altai Regional Center for the Prevention and Control of AIDS and Infectious Diseases, Barnaul
  - Regional Center for the Prevention and Control of AIDS and Infectious Diseases, Chelyabinsk
  - Center for AIDS Prevention and Control, Gorno-Altaysk
  - Center for the Prevention and Control of AIDS and Infectious Diseases, Khabarovsk
  - Clinical Center for AIDS Prevention and Control, Krasnodar
  - The State Budgetary Healthcare Institution of Moscow "Infectious Clinical Hospital No. 2 of the Moscow City Health Department" (SGBU ICD No. 2 DZM), Moscow City Center for AIDS Prevention and Control of the Moscow City Health Department, Moscow
  - State Regional Clinical Hospital "City Infectious Clinical Hospital No. 1", Novosibirsk
  - Center for AIDS Prevention and Control, Rostov-on-Don
  - State Public Health Institution of the Leningrad Region "Center for the Prevention and Control of AIDS and Infectious Diseases", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "Center for the Prevention and Control of AIDS and Infectious Diseases", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No